CLINICAL TRIAL: NCT00943228
Title: Intensified Dosing of Cellcept in Kidney Transplantation Trial
Brief Title: Intensified Dosing of Cellcept (Mycophenolate Mofetil) in Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IDOC001
Record Dates: First submitted 2009-07-06; First posted 2009-07-22 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Acute Rejection of Renal Transplant
Keywords: Renal transplantation; Adequate exposure; Acute rejection; mycophenolate mofetil; immunosuppression
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mycophenolate mofetil (Experimental): mycophenolate mofetil 2000mg BID (4g/day) for 14 days, followed by mycophenolate 1000mg BID (2g/day) thereafter
  Interventions: Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: mycophenolate mofetil — High dose 4gms daily
  Other Names: MMF; Cellcept

SUMMARY:
The primary objective of this study is to determine whether 4 grams daily of mycophenolate mofetil (MMF) results in a greater proportion of individuals adequately exposed as measured by drug levels (area under the curve of > 40 mg*hr/L).

DETAILED DESCRIPTION:
Several studies have shown that early exposure to adequate levels of immunosuppression are required to reduce acute rejection rates in kidney transplantation.(1, 2) Our center has shown that early exposure of mycophenolate mofetil (MMF or Cellcept) is associated with acute rejection rates and that many patients are underexposed in the early transplant period.(2) In a recently completed multicenter Canadian (CLEAR) study we found that higher doses of mycophenolate mofetil (MMF 3 grams daily versus 2 grams daily) were associated with better early exposure by day 5 and that this was associated with less rejection but no increase in toxicity.(3) The best cut point that discriminated between low and high rejection rates was a mycophenolic acid (MPA) 12 hour area under the curve (AUC) of 40 mg*hr/L. Patients below this level experienced rejection rates of 50% compared to <16% for those above this level. Even with the higher dose 26% of subjects were inadequately exposed. Since medication adjustments based on drug levels is hampered by steady state conditions and the turn around time of MPA testing we are interested in exploring even higher initial doses of MMF with the aim to maximize the numbers of patients achieving adequate early exposure to MPA.

Objectives:

The primary objective of this study is to determine whether 4 gms daily of MMF results in a greater proportion of individuals adequately exposed as measured by a day 5 MPA AUC of >40 mg*hr/L.

The secondary objectives of this study are to assess the ability of this strategy to achieve target MPA AUC exposure of 40-60 mg*hr/L by day 14 and to determine the distribution of MMF doses that are necessary to achieve this level of exposure. Safety data (hemoglobin and WBC counts, need for further dose changes based on gastrointestinal intolerance, acute rejection, renal function, and wound infection) will be also collected over the first 3 months post transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing single organ kidney transplantation.
* Age > 18 years old.
* Patients who would normally receive our standard therapy of basiliximab, tacrolimus, MMF and steroids.
* All patients will be required to sign informed consent.

Exclusion Criteria:

* Patients will be excluded if they require anti-thymocyte induction therapy, have documented gastroparesis, have known intolerance to MMF, or are prescribed cyclosporine.
* As a standard policy all women of childbearing age will be informed about the risks of all immunosuppressive drugs on fetal outcomes and will be required to use 2 forms of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Adequate drug exposure. MPA AUC > 40 mg*hr/l | First two weeks - 14 days

SECONDARY OUTCOMES:
Gastrointestinal symptoms (nausea, vomiting, abdominal pain, diarrhea). | First two weeks - 14 days
Leukopenia, anemia, thrombocytopenia and infection. | First two weeks - 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bryce A Kiberd, MD, Principal Investigator — Dalhousie University
Locations (1):
- QE II Health Sciences Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Kiberd BA, Lawen J, Daley C. Limits to intensified mycophenolate mofetil dosing in kidney transplantation. Ther Drug Monit. 2012 Dec;34(6):736-8. doi: 10.1097/FTD.0b013e31826d7bfa. PMID 23007746